CLINICAL TRIAL: NCT03539484
Title: A First-in-Human, Open-Label, Multicenter, Dose-Escalation Phase I Clinical Study of Single-Agent RO7172508 in Patients With Locally Advanced and/or Metastatic CEA-Positive Solid Tumors
Brief Title: A Study of RO7172508 in Patients With Locally Advanced and/or Metastatic CEA-Positive Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to change in benefit-risk ratio, driven by high incidence GI toxicity in absence of clinically significant anti-tumor efficacy.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP40092
Record Dates: First submitted 2018-04-19; First posted 2018-05-29 (Actual); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — obinutuzumab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I: Single Participant Cohorts IV/MAD-Escalation (Experimental): Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W). The starting dose of RO7172508 was 65 microgram (mcg) and the maximum dose explored was 1.6 milligram (mg).
  Interventions: Drug: RO7172508; Drug: Tocilizumab
- Part II: Multiple Participant Cohorts IV/MAD-Escalation (Experimental): Multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts: The starting-dose for the initiation of the IV dose-escalation was determined by Part I and RO7172508 was initially given Q3W. Dose-escalation was undertaken based on safety until determination of the MTD or the highest safe dose if MTD is not reached. If on-target toxicity was reported in the first cycle of treatment, fractionated dosing may be implemented for the first cycle to improve tolerability.
  Interventions: Drug: RO7172508; Drug: Obinutuzumab; Drug: Tocilizumab
- Part II: Multiple Participant Cohorts SC/MAD-Escalation (QW) (Experimental): Multiple ascending dose-escalation of SC-administered RO7172508 in multiple participant cohorts. These will be initiated once the IV schedule has shown RO7172508 preliminary clinical activity or the MTD has been established and is equal to or above 2 mg. The starting-dose and regimen once a week or once every 3 weeks (QW or Q3W) for SC administration will be proposed based on the evaluation of the safety and PK data observed following IV administration but will not exceed the highest safe dose tested in the IV Q3W dose escalation; a minimum dose of 2 mg is defined for a single SC administration. In addition, the QW SC starting-dose will not exceed one third of the IV MTD or of the highest safe IV dose tested. Dose escalation will continue based on safety until determination of the MTD or the planned maximum dose of 400 mg. If on-target toxicity is reported in the first cycle of treatment, fractionated dosing may be implemented for the first cycle to improve tolerability.
  Interventions: Drug: RO7172508; Drug: Obinutuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO7172508 — RO7172508 was administered at a dose and as per the schedule specified in the respective arms.
Drug: Obinutuzumab — In the event obinutuzumab treatment is implemented, obinutuzumab will be administered either on Day-7 or on Day-7 and Day-6. If obinutuzumab is given only on one day, then the schedule for Day-7 should be followed including an end of infusion sample.
  Arms: Part II: Multiple Participant Cohorts IV/MAD-Escalation; Part II: Multiple Participant Cohorts SC/MAD-Escalation (QW)
Drug: Tocilizumab — Tocilizumab was administered if required, for the management of severe CRS (cytokine release syndrome)

SUMMARY:
This study was to determine the maximum-tolerated dose (MTD) and/or the optimal biological dose (OBD) as well as the optimal schedule for intravenous (IV) and subcutaneous (SC) administrations of RO7172508 as monotherapy, with or without obinutuzumab pre-treatment, in participants with locally advanced and/or metastatic carcinoembryonic antigen (CEA)-positive solid tumors who have progressed on standard of care (SOC) treatment, are intolerant to SOC, and/or are non-amenable to SOC. This study was conducted in two parts. Part I of the study consisted of an IV single participant cohort/multiple-ascending dose-escalation to evaluate the safety of RO7172508. Part II was a multiple participant cohort/multiple-ascending dose-escalation to define the MTD and/or OBD of RO7172508 administered as single agent, IV and/or SC, in participants with tumors that are expressing high as well as moderate/low-CEA. The study switched from Part I to Part II when the maximum planned dose for Part I was reached or the occurrence of a RO7172508-related Grade >= 2 adverse event (AE) or dose-limiting toxicity (DLT) was observed, whichever comes first. The Sponsor may decide to switch from Part I to Part II in the absence of an observed RO7172508-related Grade >= 2 toxicity or prior to maximum planned dose for Part I.

ELIGIBILITY:
Inclusion Criteria:

* For Part I: participants with locally advanced and/or metastatic solid tumor with confirmed cytoplasmic and/or membranous high CEA expression in tumor tissue is required. Participants must have progressed on a SOC therapy, be intolerant to SOC, and/or are non-amenable to SOC.
* For <12 mg dose cohorts, serum CEA levels below a certain threshold is required as follows:

  * For dose cohorts 65-159 microgram, a sCEA level of < 22 ng/mL
  * For dose cohorts 160-399 microgram, a sCEA level of < 28 ng/mL
  * For dose cohorts 400-799 microgram, a sCEA level of < 44 ng/mL
  * For dose cohorts 800-1599 microgram, a sCEA level of < 70 ng/mL
  * For the dose cohort of 1.6-3.1 milligram, a sCEA level of < 123 ng/mL
  * For the dose cohort of 3.2-6.3 milligram, an sCEA level of < 229 ng/mL.
  * For the dose cohort of 6.4-11.9 milligram, an sCEA level of < 440 ng/mL. If dose fractionation is implemented, the sCEA threshold for inclusion should correspond to the dose range of the first dose administered.
* For Part II, participants with locally advanced and/or metastatic solid tumor expressing cytoplasmic and/or membranous high-CEA or moderate/low-CEA on archival material, who have progressed on a SOC therapy, are intolerant to SOC, and/or are non-amenable to SOC. Participants must have a lesion amenable to biopsy (except participants with NSCLC, which may be enrolled with archival tissue available only). For participants with colorectal cancer (CRC) only, the CEA assessment by immunohistochemistry should be performed but the result is not required to enroll the participant.
* Radiologically measurable disease according to RECIST v1.1.
* Life expectancy of >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade <= 1 or returned to baseline except alopecia (any grade) and Grade 2 peripheral neuropathy.
* Adequate hematological, liver, renal, and lung function
* For women: agree to remain abstinent or use two contraceptive methods that result in a failure rate of <1% per year from screening until 2 months after the last dose of RO7172508 and have a negative pregnancy test within one week prior to the first study treatment administration
* For men: remain abstinent or use contraceptive measures such as a condom plus an additional contraceptive method that together result in a failure rate of <1% per year, with partners who are woman of childbearing potential and refrain from donating sperm during the study

Exclusion Criteria:

* History or clinical evidence of central nervous system (CNS) primary tumors or metastases unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days before screening.
* Non-irradiated lesions > 2 cm at critical sites where tumor swelling induced by RO7172508 is expected to lead to significant complications.
* Another invasive malignancy in the last 2 years
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or contraindicate the use of an investigational drug.
* Uncontrolled hypertension, unstable angina, congestive heart failure, serious cardiac arrhythmia that requires treatment with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia, and history of myocardial infarction within 6 months of enrollment.
* Active or uncontrolled infections.
* Known hepatitis B or C
* Major surgery or significant traumatic injury < 28 days prior to the first RO7172508 administration or anticipation of the need for major surgery during study treatment.

Specific Exclusion Criteria if Pre-treatment with Obinutuzumab is Implemented:

* Known HIV
* Positive test results for HBV infection, HBcAb indicating an active viral infection and positive test results for HCV.
* Participants positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
* History of progressive multifocal leukoencephalopathy.
* Active TB requiring treatment within 3 years prior to baseline.
* Latent TB diagnosed during Screening.
* Positive test results for human T-lymphotropic virus 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Cliniques Universitaires St-Luc, Brussels, Belgium
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Spain (3):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- PART1 - RO7172508 - Q3W - 65 mcg: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 65 microgram (mcg).
- PART1 - RO7172508 - Q3W - 160 mcg: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 160 microgram (mcg).
- PART1 - RO7172508 - Q3W - 400 mcg: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 400 microgram (mcg).
- PART2 - RO7172508 - Q3W - 400 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts: The starting-dose for the initiation of the IV dose-escalation was determined by Part I and RO7172508 was initially given Q3W. Starting dose of RO7172508 was 400 mcg.
- PART2 - RO7172508 - Q3W - 800 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts. RO7172508 was administered intravenously at a dose of 800 mcg.
- PART2 - RO7172508 - Q3W - 1200 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts. RO7172508 was administered intravenously at a dose of 1200 mcg.
- PART2 - RO7172508 - Q3W - 1800 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts. RO7172508 was administered intravenously at a dose of 1800 mcg.
Period: Overall Study
Arm/Group | PART1 - RO7172508 - Q3W - 65 mcg | PART1 - RO7172508 - Q3W - 160 mcg | PART1 - RO7172508 - Q3W - 400 mcg | PART2 - RO7172508 - Q3W - 400 mcg | PART2 - RO7172508 - Q3W - 800 mcg | PART2 - RO7172508 - Q3W - 1200 mcg | PART2 - RO7172508 - Q3W - 1800 mcg
Started | 1 | 1 | 1 | 3 | 13 | 5 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 3 | 13 | 5 | 2
Not completed — Death | 1 | 0 | 0 | 2 | 8 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 1 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PART1 - RO7172508 - Q3W - 65 mcg | PART1 - RO7172508 - Q3W - 160 mcg | PART1 - RO7172508 - Q3W - 400 mcg | PART2 - RO7172508 - Q3W - 400 mcg | PART2 - RO7172508 - Q3W - 800 mcg | PART2 - RO7172508 - Q3W - 1200 mcg | PART2 - RO7172508 - Q3W - 1800 mcg | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (NA) — Not estimable because there was 1 participant. | 60.0 (NA) — Not estimable because there was 1 participant. | 60.0 (NA) — Not estimable because there was 1 participant. | 53.7 (9.6) | 62.2 (9.0) | 58.8 (13.5) | 55.5 (16.3) | 59.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 7 | 4 | 2 | 14
  Male | 1 | 1 | 1 | 2 | 6 | 1 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 3 | 13 | 5 | 2 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 3 | 13 | 5 | 2 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Number of participants with DLTs.
Time Frame: Up to approximately 12 months
Population: DLT evaluble population included participants who completed the DLT window without a DLT, or participants who reported with a DLT.
Measure: Number; unit: Participants
Groups:
- Part I: Single Participant Cohort IV RO7172508 65 mcg: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 65 microgram (mcg).
- Part I: Single Participant Cohort IV RO7172508 160 mcg: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 160 microgram (mcg).
- Part I: Single Participant Cohort IV RO7172508 400 mcg: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 400 microgram (mcg).
- Part II: Multiple Participant Cohorts IV 400 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts: The starting-dose for the initiation of the IV dose-escalation was determined by Part I and RO7172508 was initially given Q3W. Starting dose of RO7172508 was 400 mcg.
- Part II: Multiple Participant Cohorts IV 800 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts. RO7172508 was administered intravenously at a dose of 800 mcg.
- Part II: Multiple Participant Cohorts IV 1200 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts. RO7172508 was administered intravenously at a dose of 1200 mcg.
- Part II: Multiple Participant Cohorts IV 1800 mcg: Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts. RO7172508 was administered intravenously at a dose of 1800 mcg.
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 13 | 5 | 2
Participants |  |  | 0 | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Part I: Single Participant Cohort IV RO7172508 400 mcg vs Part II: Multiple Participant Cohorts IV 400 mcg vs Part II: Multiple Participant Cohorts IV 800 mcg vs Part II: Multiple Participant Cohorts IV 1200 mcg vs Part II: Multiple Participant Cohorts IV 1800 mcg; Test type: Other — A Bayesian approach is used to estimate the maximum tolerated dose (MTD); Regression, Logistic — There is no p-value derived; logistic regression is used to estimate the probability of DLT; Posterior probability at dose 1.8 mg = 10.6, 95% CI 2-sided [2.10 to 26.5]

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with adverse events.
Time Frame: 60 days after last dose of study treatment (up to approximately 12 months)
Population: Safety population included all participants enrolled in the study who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100

3. Secondary Outcome: Maximum Concentration of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: Pharmacokinetic population included all participants who received at least one dose of study treatment and who had data from at least one post-dose sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part I and Part II: Participant Cohorts IV 400 mcg: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 400 microgram (mcg). Part II was a multiple ascending dose-escalation of IV-administered RO7172508 in multiple participant cohorts: The starting-dose for the initiation of the IV dose-escalation was determined by Part I and RO7172508 was initially given Q3W. Starting dose of RO7172508 was 400 mcg.
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 4 | 13 | 5 | 2
ng/mL
  Baseline sCEA <=20 ng/mL: number analyzed (Participants) | 1 | 1 | 2 | 6 | 3 | 1
  Baseline sCEA <=20 ng/mL | 9.19 | 21.5 | 73.3 (54.4) | 252 (138) | 370 (29.2) | 937
  Baseline sCEA >20 ng/mL: number analyzed (Participants) | 0 | 0 | 2 | 7 | 2 | 1
  Baseline sCEA >20 ng/mL |  |  | 85.0 (17.3) | 184 (167) | 290 (2.9) | 1180

4. Secondary Outcome: Time of Maximum Concentration of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: as for outcome 3
Measure: Median (Full Range); unit: Hour
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 4 | 13 | 5 | 2
Hour
  Baseline sCEA <=20 ng/mL: number analyzed (Participants) | 1 | 1 | 2 | 6 | 3 | 1
  Baseline sCEA <=20 ng/mL | 2.58 | 2.07 | 3.30 [2.20 to 4.40] | 3.79 [1.80 to 4.10] | 2.13 [2.10 to 3.80] | 4.48
  Baseline sCEA >20 ng/mL: number analyzed (Participants) | 0 | 0 | 2 | 7 | 2 | 1
  Baseline sCEA >20 ng/mL |  |  | 2.16 [2.16 to 2.16] | 2.18 [2.00 to 4.30] | 3.09 [2.00 to 4.20] | 1.95

5. Secondary Outcome: Clearance or Apparent Clearance of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 3 | 8 | 4 | 2
mL/hr
  Baseline sCEA <=20 ng/mL: number analyzed (Participants) | 1 | 1 | 2 | 5 | 3 | 1
  Baseline sCEA <=20 ng/mL | 332 | NA — Not determined because λz was not estimable. | 111 (34.4) | 55.4 (61.5) | 67.4 (49.2) | 34.8
  Baseline sCEA >20 ng/mL: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 1
  Baseline sCEA >20 ng/mL |  |  | 453 | 340 (527) | 68.8 | 39.3

6. Secondary Outcome: Volume of Distribution at Steady State of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: Analysis not conducted due to participants not reaching steady state due to early withdrawal or loss of exposure due to immunogenicity.
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Plasma Concentration Time-Curve From Zero to the Last Measured Concentration (AUClast) of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 4 | 13 | 5 | 2
day*ng/mL
  Baseline sCEA <=20 ng/mL: number analyzed (Participants) | 1 | 1 | 2 | 6 | 3 | 1
  Baseline sCEA <=20 ng/mL | 6.93 | 1.91 | 143 (38.4) | 411 (137) | 740 (49.4) | 2140
  Baseline sCEA >20 ng/mL: number analyzed (Participants) | 0 | 0 | 2 | 7 | 2 | 1
  Baseline sCEA >20 ng/mL |  |  | 45.4 (34.4) | 83.5 (178) | 370 (121) | 1910

8. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve Computed From Time of Dosing to Infinity (AUCinf) of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 3 | 8 | 4 | 2
day*ng/mL
  Baseline sCEA <=20 ng/mL: number analyzed (Participants) | 1 | 1 | 2 | 5 | 3 | 1
  Baseline sCEA <=20 ng/mL | 8.15 | NA — Not determined because λz was not estimable. | 150 (34.7) | 602 (61.7) | 740 (49.2) | 2160
  Baseline sCEA >20 ng/mL: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 1
  Baseline sCEA >20 ng/mL |  |  | 36.8 | 98.1 (527) | 727 | 1910

9. Secondary Outcome: Dose Normalized Area Under the Serum Concentration Versus Time Curve Computed From Time of Dosing to Infinity (AUCinf/Dose) of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 3 | 8 | 4 | 2
day*ng/mL
  Baseline sCEA <=20 ng/mL: number analyzed (Participants) | 1 | 1 | 2 | 5 | 3 | 1
  Baseline sCEA <=20 ng/mL | 125 | NA — Not determined because λz was not estimable. | 375 (34.2) | 753 (61.6) | 618 (49.3) | 1200
  Baseline sCEA >20 ng/mL: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 1
  Baseline sCEA >20 ng/mL |  |  | 92.0 | 122 (526) | 606 | 1060

10. Secondary Outcome: Half-Life of RO7172508
Time Frame: Cycle 1 following single dose administration of RO7172508
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I and Part II: Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 3 | 8 | 4 | 2
Hour
  Baseline sCEA <=20 ng/mL: number analyzed (Participants) | 1 | 1 | 2 | 5 | 3 | 1
  Baseline sCEA <=20 ng/mL | 17.1 | NA — Not determined because λz was not estimable. | 54.0 (112) | 62.1 (42.4) | 40.9 (68.9) | 48.7
  Baseline sCEA >20 ng/mL: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 1
  Baseline sCEA >20 ng/mL |  |  | 9.27 | 22.0 (43.9) | 23.3 | 18.4

11. Secondary Outcome: Presence or Absence and Titer of ADAs
Time Frame: Up to approximately 12 months
Population: Participants were considered as evaluable for immunogenicity analysis if they had at least 3 cycles of treatment to allow for development of potential ADAs.
Measure: Number; unit: Participants
Groups:
- Part I: Single Participant Cohort IV RO7172508 65 mcgEdit: Part I was a multiple-ascending dose-escalation in single participant cohorts. RO7172508 was administered intravenously once every 3 weeks (Q3W) at a dose of 65 microgram (mcg).
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcgEdit | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Participants
  Presence of ADAs | 0 | 0 | 1 | 3 | 5 | 2 | 0
  Positive Titer | 0 | 0 | 1 | 3 | 5 | 2 | 0

12. Secondary Outcome: Changes in Frequency of Tumor Infiltrating Lymphocytes
Time Frame: Cycle 1 Day 1 (Pre-treatment), Cycle 2 Day 8 (Cycle is 21 days)
Population: Biopsies were not mandatory in part 1. Results from 2 participants are excluded as measured using a different assay.
Measure: Median (Full Range); unit: % of CD3
Units Other Than Participants: Results
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 3 | 0
% of CD3
  CD8 TIL Pre-treatment (Cycle 1 Day 1): number analyzed (Results) | 0 | 0 | 0 | 1 | 9 | 3 | 0
  CD8 TIL Pre-treatment (Cycle 1 Day 1) |  |  |  | 48.2 [48.2 to 48.2] | 41.40 [29.5 to 75.6] | 64.4 [40.0 to 68.2] |
  CD8 TIL On-treatment (Cycle 2 Day 8): number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 2 | 0
  CD8 TIL On-treatment (Cycle 2 Day 8) |  |  |  | 54.15 [51.2 to 57.1] | 54.7 [38.0 to 78.4] | 52.75 [35.4 to 70.1] |
  CD4 TIL Pre-treatment (Cycle 1 Day 1): number analyzed (Results) | 0 | 0 | 0 | 1 | 9 | 3 | 0
  CD4 TIL Pre-treatment (Cycle 1 Day 1) |  |  |  | 39.7 [39.7 to 39.7] | 35.70 [15.3 to 60.3] | 22.90 [22.5 to 58.2] |
  CD4 TIL On-treatment (Cycle 2 Day 8): number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 2 | 0
  CD4 TIL On-treatment (Cycle 2 Day 8) |  |  |  | 35.00 [32.8 to 37.2] | 33.80 [2.4 to 54.9] | 42.65 [29.9 to 55.4] |

13. Secondary Outcome: Secondary: Changes in Activation Status of Tumor Infiltrating Lymphocytes (% of CD8)
Time Frame: Cycle 1 Day 1 (Pre-treatment), Cycle 2 Day 8 (Cycle is 21 days)
Population: Biopsies were not mandatory in part 1. Results from 2 participants are excluded as measured using a different assay.
Measure: Median (Full Range); unit: % of CD8
Units Other Than Participants: Results
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 3 | 0
% of CD8
  CD8+CD25+ Pre-treatment (Cycle 1 Day 1): number analyzed (Results) | 0 | 0 | 0 | 1 | 9 | 3 | 0
  CD8+CD25+ Pre-treatment (Cycle 1 Day 1) |  |  |  | 22.00 [22.0 to 22.0] | 17.60 [3.3 to 89.9] | 9.70 [9.1 to 29.5] |
  CD8+CD25+ On-treatment (Cycle 2 Day 8): number analyzed (Results) | 0 | 0 | 0 | 2 | 8 | 2 | 0
  CD8+CD25+ On-treatment (Cycle 2 Day 8) |  |  |  | 25.80 [25.4 to 26.2] | 35.30 [3.7 to 57.7] | 19.60 [13.1 to 26.1] |
  CD8+CD279+ Pre-treatment (Cycle 1 Day 1): number analyzed (Results) | 0 | 0 | 0 | 1 | 9 | 3 | 0
  CD8+CD279+ Pre-treatment (Cycle 1 Day 1) |  |  |  | 11.90 [11.9 to 11.9] | 8.70 [2.3 to 70.8] | 11.40 [6.2 to 72.3] |
  CD8+CD279+ On-treatment (Cycle 2 Day 8): number analyzed (Results) | 0 | 0 | 0 | 2 | 8 | 2 | 0
  CD8+CD279+ On-treatment (Cycle 2 Day 8) |  |  |  | 16.80 [13.0 to 20.6] | 23.20 [7.5 to 76.7] | 7.90 [4.3 to 11.5] |

14. Secondary Outcome: Changes in Activation Status of Tumor Infiltrating Lymphocytes (% of CD4)
Time Frame: Cycle 1 Day 1 (Pre-treatment), Cycle 2 Day 8 (Cycle is 21 days)
Population: Biopsies were not mandatory in part 1. Results from 2 participants are excluded as measured using a different assay.
Measure: Median (Full Range); unit: % of CD4
Units Other Than Participants: Results
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 3 | 0
% of CD4
  CD4+CD25+ Pre-treatment (Cycle 1 Day 1): number analyzed (Results) | 0 | 0 | 0 | 1 | 9 | 3 | 0
  CD4+CD25+ Pre-treatment (Cycle 1 Day 1) |  |  |  | 51.9 [51.9 to 51.9] | 41.20 [11.4 to 86.8] | 26.90 [20.6 to 34.4] |
  CD4+CD25+ On-treatment (Cycle 2 Day 8): number analyzed (Results) | 0 | 0 | 0 | 2 | 6 | 2 | 0
  CD4+CD25+ On-treatment (Cycle 2 Day 8) |  |  |  | 47.35 [42.3 to 52.4] | 47.65 [12.0 to 51.8] | 30.75 [11.5 to 50.0] |
  CD4+CD279+ Pre-treatment (Cycle 1 Day 1): number analyzed (Results) | 0 | 0 | 0 | 1 | 9 | 3 | 0
  CD4+CD279+ Pre-treatment (Cycle 1 Day 1) |  |  |  | 16.50 [16.5 to 16.5] | 10.90 [1.8 to 43.8] | 16.80 [4.0 to 32.8] |
  CD4+CD279+ On-treatment (Cycle 2 Day 8): number analyzed (Results) | 0 | 0 | 0 | 2 | 6 | 2 | 0
  CD4+CD279+ On-treatment (Cycle 2 Day 8) |  |  |  | 27.40 [18.7 to 36.1] | 24.30 [12.0 to 58.7] | 22.40 [11.5 to 33.3] |

15. Secondary Outcome: Changes in Spatial Distribution of Tumor Infiltrating Lymphocytes
Description: Spatial distribution of TIL's analyzed by performing IHC assay, which measures the density and intra-tumoral location of CD8+ T cells and reports "CD8 T cell immune phenotypes". These are classified as "desert", "excluded" and "inflamed".
Time Frame: Cycle 1 Day 1 (Pre-treatment), Cycle 2 Day 8 (Cycle is 21 days)
Population: Paired included participant's with different dose and actual exposure levels. Data were pooled across all dose levels because the number of biopsy evaluable participants was overall small, and no dose/response relationship was found.
Measure: Number; unit: CD8 immune phenotype
Units Other Than Participants: Results
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 4 | 2
CD8 immune phenotype
  Pre-treatment (Cycle 1 Day 1) Desert: number analyzed (Results) | 0 | 0 | 0 | 1 | 7 | 2 | 2
  Pre-treatment (Cycle 1 Day 1) Desert |  |  |  | 1 | 5 | 0 | 0
  Pre-treatment (Cycle 1 Day 1) Excluded: number analyzed (Results) | 0 | 0 | 0 | 1 | 7 | 2 | 2
  Pre-treatment (Cycle 1 Day 1) Excluded |  |  |  | 0 | 0 | 1 | 1
  Pre-treatment (Cycle 1 Day 1) Inflamed: number analyzed (Results) | 0 | 0 | 0 | 1 | 7 | 2 | 2
  Pre-treatment (Cycle 1 Day 1) Inflamed |  |  |  | 0 | 2 | 1 | 1
  On-treatment (Cycle 2 Day 8) Desert: number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 4 | 0
  On-treatment (Cycle 2 Day 8) Desert |  |  |  | 2 | 6 | 1 |
  On-treatment (Cycle 2 Day 8) Excluded: number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 4 | 0
  On-treatment (Cycle 2 Day 8) Excluded |  |  |  | 0 | 1 | 2 |
  On-treatment (Cycle 2 Day 8) Inflamed: number analyzed (Results) | 0 | 0 | 0 | 2 | 9 | 4 | 0
  On-treatment (Cycle 2 Day 8) Inflamed |  |  |  | 0 | 2 | 1 |

16. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response was defined as a Complete Response (CR) or Parital Response (PR), as determined by the Investigator's assessment using RECIST v1.1 and confirmed by repeat assessments >= 4 weeks after initial documentation. To classify a response as SD, measurements are classified as stable (according to RECIST v1.1) at least once after study entry at a minimum of 6 weeks after study entry.
Time Frame: Up to approximately 12 months
Population: Efficacy population included all participants who received at least one dose of RO7172508.
Measure: Number; unit: Participants
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is determined as the rate of participants with an observed tumor response of CR or PR (ORR) or CR, PR or SD (DCR). DCR is to be derived for RECIST v1.1.
Time Frame: Up to approximately 12 months
Population: Efficacy population included all participants who received at least one dose of RO7172508.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 13 | 5 | 2
Participants | 0 | 0 | 0 | 1 | 3 | 1 | 0

18. Secondary Outcome: Duration of Response (DOR)
Description: Among participants with an objective response (responders), DOR will be defined as the time from first occurrence of a documented objective response until the time of documented disease progression or death within 30 days from last study treatment from any cause during treatment, whichever occurs first. This will be calculated for participants who have a best overall response of CR or PR as defined per RECIST v1.1 and per iRECIST.
Time Frame: Up to approximately 12 month
Population: Efficacy population included all participants who received at least one dose of RO7172508. DOR was not calculated because none of the participants had a response (complete or partial).
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS (on-treatment) will be defined as the time from study treatment initiation (Cycle 1 Day 1) to the first occurrence of documented disease progression or death from any cause during treatment (death within 30 days from last study treatment), whichever occurs first.
Time Frame: Up to approxmately 12 months
Population: Efficacy population included all participants who received at least one dose of RO7172508. PFS was not calculated because number of evaluable participants in each cohort respectively was too small to obtain reliable estimates for this endpoint.
Arm/Group | Part I: Single Participant Cohort IV RO7172508 65 mcg | Part I: Single Participant Cohort IV RO7172508 160 mcg | Part I: Single Participant Cohort IV RO7172508 400 mcg | Part II: Multiple Participant Cohorts IV 400 mcg | Part II: Multiple Participant Cohorts IV 800 mcg | Part II: Multiple Participant Cohorts IV 1200 mcg | Part II: Multiple Participant Cohorts IV 1800 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 12 months
Description: The safety population included all participants enrolled in the study who received at least one dose of study treatment.
Arm/Group | PART1 - RO7172508 - Q3W - 65 mcg | PART1 - RO7172508 - Q3W - 160 mcg | PART1 - RO7172508 - Q3W - 400 mcg | PART2 - RO7172508 - Q3W - 400 mcg | PART2 - RO7172508 - Q3W - 800 mcg | PART2 - RO7172508 - Q3W - 1200 mcg | PART2 - RO7172508 - Q3W - 1800 mcg
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 2/3 | 8/13 | 3/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/1 | 0/3 | 8/13 | 3/5 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 3/3 | 13/13 | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PART1 - RO7172508 - Q3W - 65 mcg (N=1) | PART1 - RO7172508 - Q3W - 160 mcg (N=1) | PART1 - RO7172508 - Q3W - 400 mcg (N=1) | PART2 - RO7172508 - Q3W - 400 mcg (N=3) | PART2 - RO7172508 - Q3W - 800 mcg (N=13) | PART2 - RO7172508 - Q3W - 1200 mcg (N=5) | PART2 - RO7172508 - Q3W - 1800 mcg (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PART1 - RO7172508 - Q3W - 65 mcg (N=1) | PART1 - RO7172508 - Q3W - 160 mcg (N=1) | PART1 - RO7172508 - Q3W - 400 mcg (N=1) | PART2 - RO7172508 - Q3W - 400 mcg (N=3) | PART2 - RO7172508 - Q3W - 800 mcg (N=13) | PART2 - RO7172508 - Q3W - 1200 mcg (N=5) | PART2 - RO7172508 - Q3W - 1800 mcg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (12) | 2 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye haematoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 1 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (6) | 3 (5) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 3 (6) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 3 (8) | 3 (11) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 4 (5) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Intercepted medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 5 (5) | 3 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (2) | 1 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
RO7172508 SC not initiated; max tolerated dose IV below starting dose for SC. Study terminated due to change in benefit-risk ratio, driven by high incidence GI toxicity in absence of clinically significant anti-tumor efficacy at dose levels tested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT03539484/Prot_SAP_000.pdf